CLINICAL TRIAL: NCT00886236
Title: The Effect of Gabapentin on Acute Pain and PONV in Bariatric Surgical Patients
Brief Title: Study of the Effect of the Drug Gabapentin on Postoperative Pain and Incidence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR # 18041 Gaba Bariatric
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Obesity, Morbid; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Gastric Bypass; Gabapentin; Postoperative Nausea and Vomiting; Analgesics, Opioids; Sleep Apnea, Obstructive; Respiratory Depression; Oximetry
MeSH Terms: conditions — Obesity, Morbid; Pain, Postoperative; Postoperative Nausea and Vomiting; Sleep Apnea, Obstructive; Respiratory Insufficiency | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Preoperative Gabapentin Liquid (Active Comparator): Preoperative Gabapentin Elixir (1200 mg) AND Postoperative Placebo Elixir (300 mg x 6 doses)
  Interventions: Drug: Gabapentin
- 2 Preoperative and Postoperative Gabapentin Liquid (Experimental): Preoperative Gabapentin Elixir (1200 mg) AND Postoperative Gabapentin Elixir (300 mg x 6 doses)
  Interventions: Drug: Gabapentin
- 3 Preoperative and Postoperative Placebo Liquid (Placebo Comparator): Preoperative Placebo Liquid (1200 mg) AND Postoperative Placebo Elixir (300 mg x 6 doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 1200 mg (24 cc) by mouth 1 hour prior to surgery AND Gabapentin 300 mg (6cc) by mouth x 6 doses after surgery (0800PM the evening of surgery, 0800AM postoperative day 1, 0200PM postoperative day 1, 0800PM postoperative day 1, 0800AM postoperative day 2, 1200PM postoperative day 2)
  Arms: 2 Preoperative and Postoperative Gabapentin Liquid
Drug: Placebo — Placebo 1200 mg (24 cc) by mouth 1 hour prior to surgery AND Placebo 300 mg (6cc) by mouth x 6 doses after surgery (0800PM the evening of surgery, 0800AM postoperative day 1, 0200PM postoperative day 1, 0800PM postoperative day 1, 0800AM postoperative day 2, 1200PM postoperative day 2)
  Arms: 3 Preoperative and Postoperative Placebo Liquid
Drug: Gabapentin — Gabapentin 1200 mg (24 cc) by mouth 1 hour prior to surgery AND Placebo 300 mg (6cc) by mouth x 6 doses after surgery (0800PM the evening of surgery, 0800AM postoperative day 1, 0200PM postoperative day 1, 0800PM postoperative day 1, 0800AM postoperative day 2, 1200PM postoperative day 2)
  Arms: 1 Preoperative Gabapentin Liquid

SUMMARY:
The purpose of this research study is to evaluate the drug gabapentin (Neurontin®) for its ability to reduce postoperative pain, the need for morphine-like pain medication, and the severity and frequency of postoperative nausea and vomiting in laparoscopic gastric bypass surgery patients.

DETAILED DESCRIPTION:
The occurrence of morbid obesity is at epidemic proportions in the United States. Laparoscopic gastric bypass is an effective means of safely facilitating patient weight loss and thereby drastically reducing the prevalence and severity of many future health complications [1]. However, managing morbidly obese surgical patients poses certain obstacles for anesthesiologists, including a high incidence of obstructive sleep apnea [2].

Laparoscopic gastric bypass, like all surgical interventions, has associated postoperative challenges including pain management and prevention/control of postoperative nausea and vomiting. To assure the highest patient satisfaction, all areas of patient comfort must be addressed. However, with pain management in morbidly obese patients, caution must be used when administering opioids, as they can have an increasing effect of respiratory depression in patients already at risk due to obstructive sleep apnea [3]. Gastric bypass is also associated with a significant incidence of protracted postoperative nausea and vomiting [4]. Therefore, regimens that address both patient safety and patient comfort are desired.

Gabapentin (Neurontin) is an alkylated analog of the inhibitory neurotransmitter gamma-aminobutyric acid (GABA) that has been FDA approved for the treatment of seizures, headaches fibromyalgia and chronic neuropathic pain due to various etiologies [5]. Many randomized controlled trials have been performed with perioperative gabapentin [6-10]. The effect of perioperative administration of gabapentin on postoperative pain and opioid consumption has been extensively studied and several meta-analyses have been published in the last several years examining to overall findings of these studies. The general consensus is that gabapentin has anti-hyperalgesic and opioid-sparing properties and may also reduce the incidence of postoperative nausea and vomiting [5, 11-15]. Most research has shown that gabapentin is beneficial in the treatment of postoperative pain, but some show neither positive nor negative effects. There has been no evidence that gabapentin is detrimental or poses any risks to the postoperative patient. However, gabapentin has not been specifically studied in bariatric surgery. Therefore, the purpose of this study is to explore the hypothesis that perioperative gabapentin has anti-hyperalgesic and opioid-sparing properties, thus increase patient comfort and satisfaction by decreasing pain scores and reducing the adverse effects of opioids, such as postoperative nausea and vomiting.

This is a randomized, double-blind and placebo controlled study, which will be performed in adult laparoscopic gastric bypass patients coming to surgery for morbid obesity. The major end-points of analyses are intraoperative and postoperative opioid requirements and the incidence of nausea and vomiting in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic gastric bypass surgery
* Age > 18 years

Exclusion Criteria:

* Patients under the age of 18 years
* Patients who undergo open gastric bypass
* Patients with a history of chronic pain treated with pregabalin, gabapentin or opioids
* Patients with a history of chronic renal disease (creatinine > 1.3)
* Patients with a history of bleeding gastric ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D McEvoy, MD, Principal Investigator — Medical University of South Carolina; Scott T Reeves, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Sowemimo OA, Yood SM, Courtney J, Moore J, Huang M, Ross R, McMillian U, Ojo P, Reinhold RB. Natural history of morbid obesity without surgical intervention. Surg Obes Relat Dis. 2007 Jan-Feb;3(1):73-7; discussion 77. doi: 10.1016/j.soard.2006.10.017. Epub 2006 Dec 27. PMID 17196439
- [Background] Feld JM, Hoffman WE, Stechert MM, Hoffman IW, Ananda RC. Fentanyl or dexmedetomidine combined with desflurane for bariatric surgery. J Clin Anesth. 2006 Feb;18(1):24-8. doi: 10.1016/j.jclinane.2005.05.009. PMID 16517328
- [Background] Kong VK, Irwin MG. Gabapentin: a multimodal perioperative drug? Br J Anaesth. 2007 Dec;99(6):775-86. doi: 10.1093/bja/aem316. PMID 18006529
- [Background] Hofer RE, Sprung J, Sarr MG, Wedel DJ. Anesthesia for a patient with morbid obesity using dexmedetomidine without narcotics. Can J Anaesth. 2005 Feb;52(2):176-80. doi: 10.1007/BF03027725. PMID 15684259
- [Background] Moussa AA, Oregan PJ. Prevention of postoperative nausea and vomiting in patients undergoing laparoscopic bariatric surgery--granisetron alone vs granisetron combined with dexamethasone/droperidol. Middle East J Anaesthesiol. 2007 Jun;19(2):357-67. PMID 17684876
- [Background] Turan A, Karamanlioglu B, Memis D, Usar P, Pamukcu Z, Ture M. The analgesic effects of gabapentin after total abdominal hysterectomy. Anesth Analg. 2004 May;98(5):1370-3, table of contents. doi: 10.1213/01.ane.0000108964.70485.b2. PMID 15105217
- [Background] Prabhakar H, Arora R, Bithal PK, Rath GP, Dash HH. The analgesic effects of preemptive gabapentin in patients undergoing surgery for brachial plexus injury--a preliminary study. J Neurosurg Anesthesiol. 2007 Oct;19(4):235-8. doi: 10.1097/ANA.0b013e3181271863. PMID 17893574
- [Background] Pandey CK, Navkar DV, Giri PJ, Raza M, Behari S, Singh RB, Singh U, Singh PK. Evaluation of the optimal preemptive dose of gabapentin for postoperative pain relief after lumbar diskectomy: a randomized, double-blind, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Apr;17(2):65-8. doi: 10.1097/01.ana.0000151407.62650.51. PMID 15840990
- [Background] Fassoulaki A, Melemeni A, Stamatakis E, Petropoulos G, Sarantopoulos C. A combination of gabapentin and local anaesthetics attenuates acute and late pain after abdominal hysterectomy. Eur J Anaesthesiol. 2007 Jun;24(6):521-8. doi: 10.1017/S0265021506002134. Epub 2007 Jan 8. PMID 17207299
- [Background] Radhakrishnan M, Bithal PK, Chaturvedi A. Effect of preemptive gabapentin on postoperative pain relief and morphine consumption following lumbar laminectomy and discectomy: a randomized, double-blinded, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Jul;17(3):125-8. doi: 10.1097/01.ana.0000167147.90544.ab. PMID 16037731
- [Background] Mathiesen O, Moiniche S, Dahl JB. Gabapentin and postoperative pain: a qualitative and quantitative systematic review, with focus on procedure. BMC Anesthesiol. 2007 Jul 7;7:6. doi: 10.1186/1471-2253-7-6. PMID 17617920
- [Background] Ho KY, Gan TJ, Habib AS. Gabapentin and postoperative pain--a systematic review of randomized controlled trials. Pain. 2006 Dec 15;126(1-3):91-101. doi: 10.1016/j.pain.2006.06.018. Epub 2006 Jul 18. PMID 16846695
- [Background] Hurley RW, Cohen SP, Williams KA, Rowlingson AJ, Wu CL. The analgesic effects of perioperative gabapentin on postoperative pain: a meta-analysis. Reg Anesth Pain Med. 2006 May-Jun;31(3):237-47. doi: 10.1016/j.rapm.2006.01.005. PMID 16701190
- [Background] Seib RK, Paul JE. Preoperative gabapentin for postoperative analgesia: a meta-analysis. Can J Anaesth. 2006 May;53(5):461-9. doi: 10.1007/BF03022618. PMID 16636030
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid
Started | 20 | 21 | 21
Completed | 18 | 17 | 17
Not Completed | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 19 | 59
  >=65 years | 0 | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 47 [30 to 64] | 47 [22 to 67] | 46 [24 to 75] | 47 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 18 | 51
  Male | 3 | 5 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Amount of Diluadid Given Postoperatively
Description: The amount of intraoperative and postoperative opioids used will be collected and analyzed for the three different arms.
Time Frame: 120 hours
Measure: Mean (Full Range); unit: ml
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid
Number analyzed (Participants) | 20 | 21 | 21
ml | 11.035 [0.4 to 28.7] | 8.7 [1.0 to 30.6] | 12.4 [0.9 to 30.6]

2. Primary Outcome: Number of Participants Who Experience Incidence of Postoperative Nausea.
Time Frame: 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid
Number analyzed (Participants) | 20 | 21 | 21
Participants | 12 | 11 | 12

3. Secondary Outcome: Evaluate Incidence of Respiratory Depression as Evidenced by Pulse Oximetry Data
Time Frame: 48 hours
Measure: Mean (Full Range); unit: % oxygen saturation
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid
Number analyzed (Participants) | 20 | 21 | 21
% oxygen saturation | 93 [69 to 97] | 94 [88 to 100] | 95 [88 to 98]

ADVERSE EVENTS:
Time Frame: Patients were followed up to 120 hours or 5 days postoperatively.
Arm/Group | 1 Preoperative Gabapentin Liquid | 2 Preoperative and Postoperative Gabapentin Liquid | 3 Preoperative and Postoperative Placebo Liquid
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes